CLINICAL TRIAL: NCT06144515
Title: Collection of Samples of Bone Marrow Aspiration From Patients With Myelodysplastic Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MNV-007
Record Dates: First submitted 2023-10-29; First posted 2023-11-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Mitochondrial; Research
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Collection of Samples of Bone Marrow Aspiration From Patients With Myelodysplastic Syndrome
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Blood is collected in order to perform in vitro research:
  1. If a routine blood test is performed for clinical tests, the sponsor will receive the results of the Complete blood count (CBC) and an additional blood sample from the same puncture of 20ml to maximum 40ml will be collected for this study.
  2. If no routine blood test is performed for clinical tests, a CBC will be performed for the study and an additional blood sample of 20ml to maximum 40ml will be collected.
  Additional Bone marrow (BM) material will be obtained from the same puncture performed for routine clinical tests:

SUMMARY:
The study Objective is to collect samples of bone marrow aspirates and peripheral blood of patients with MDS for use in non-clinical research to investigate mitochondrial function sequence and effect of mitochondrial augmentation.

DETAILED DESCRIPTION:
Mitochondrial dysfunction is often associated with MDS. Studies have shown mitochondrial DNA (mtDNA) mutations in different MDS subtypes; however, their role in the pathogenesis and disease progression are not yet clear. Point mutations were found in various locations in the mitochondrial genome including tRNAs, rRNAs, and mitochondrial proteins.

Mitochondrial fragmentation in hematopoietic stem and progenitor cells (HSPC) can lead to ineffective hematopoiesis in MDS, suggesting mitochondria as a therapeutic target for treating MDS.

Mitochondria augmentation therapy (MAT) is a novel cell technology where hematopoietic stem and progenitor cells (HSPCs) are augmented ex vivo with mitochondria obtained from donor cells or tissue. MAT is based on the demonstrated ability of isolated mitochondria to enter cells and impact mitochondrial function and metabolic activity in the recipient cells. The transfer of mitochondria from cell to cell has been demonstrated using extracellular vesicles, nanotubes, and micropinocytosis. Mitochondria entering cells provide copies of normal mtDNA, which can be further propagated via replication within the recipient cell and via intercellular transfer.

Research will include in vitro and in vivo studies with the bone marrow sample, including, among other, the following: mitochondrial augmentation of bone marrow aspiration and/or subpopulations of cells (e.g. CD34+) isolated from the bone marrow aspiration; differentiation of augmented and/or non-augmented bone marrow aspiration and/or subpopulations of cells into hematopoietic lineages (e.g. erythroid, megakaryocyte, etc); assays of mitochondrial content and function; assays of hematopoietic lineages; culture of augmented and/or non-augmented bone marrow aspiration and/or subpopulations; cryopreservation of augmented and/or non-augmented bone marrow aspiration and/or subpopulations; sequencing of mitochondrial DNA and nuclear DNA; in vivo studies of engraftment, biodistribution and function of augmented and/or non-augmented bone marrow aspiration and/or subpopulations of cells isolated from the bone marrow aspiration.

Research will include in vitro studies with the peripheral blood sample, including, among other, the following: immunophenotyping of peripheral blood cells and immune-related functional assays; mitochondrial content and function of peripheral blood cells.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of 18 years old and up.
2. Suspected or previously diagnosed with Myelodysplastic Syndrome.
3. Patient able to understand and provide voluntary written informed consent.

Exclusion Criteria:

1. History of prior allogeneic hematopoietic stem cell transplantation, cell therapy, gene therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients of 18 years old and up and suspected or previously diagnosed with Myelodysplastic Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Investigate mitochondrial content and function in MDS patient-derived cells | 1 Year
  assays of mitochondrial content and function on whole bone marrow and HSPCs assays of hematopoietic lineages;
investigate effect of mitochondrial augmentation on MDS patient-derived cells | 1 Year
  in vivo studies of engraftment, biodistribution and function of augmented and/or non-augmented bone marrow aspiration and/or subpopulations of cells isolated from the bone marrow aspiration., in vitro ability to differentiate to various hematopoeitic lineages, immunophenotyping and single cells studies of cells post-augmentation and post-differentiation
Persistence of exogenous mtDNA after mitochondrial augmentation | 1 year
  Persistence of exogenous mtDNA after in vitro or in vivo culturing

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: No